CLINICAL TRIAL: NCT05306626
Title: Building Emotion Awareness and Mental Health (BEAM): Randomized Controlled Trial for Mothers of Children 18-36 Months
Brief Title: Building Emotion Awareness and Mental Health (BEAM): Mothers of Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: University of Calgary (Other); Tactica Interactive (Unknown); Centre for Healthcare Innovation (Unknown); Research Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEAM toddler RCT
Record Dates: First submitted 2022-02-17; First posted 2022-04-01 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-03

CONDITIONS: Depression, Anxiety
Keywords: Mental health; Parenting; Maternal; Psychoeducation; E-health
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being | interventions — Mental Health

STUDY DESIGN:
Intervention Model Description: The randomized controlled trial will include two arms. For the experimental arm, 70 participants will be enrolled in the BEAM group. Participants randomized to the BEAM intervention group will receive the app-based and group telehealth BEAM program. The other 70 participants will be randomized to the control group and will receive treatment as usual. Randomization will be stratified based on which telehealth group timeslots participants identify being available for during eligibility screening.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The BEAM program group (Experimental): The BEAM Program is delivered via mobile application and weekly group telehealth sessions. BEAM includes approximately 20 minutes of weekly asynchronous video modules on parenting and mental health. Mental Health videos will provide information and emotion-regulation strategies that draw from the Unified Protocol, an evidence-based treatment for depression and anxiety disorders. Self-compassion and effective communication will also be central focuses of the mental health content. Supportive parenting videos will provide parents with emotion-focused parenting strategies and help parents understand and respond to their children's challenging emotions and behaviours. The weekly group telehealth sessions will allow participants to discuss content and ask questions, with the purpose of increasing a sense of community and social support. The online community forum will provide a space for participants to reflect on their learned skills and connect with other participants in the program.
  Interventions: Behavioral: Building Emotion Awareness and Mental Health (BEAM)
- Treatment as usual group (No Intervention): The treatment as usual (TAU) control arm of the study is designed to account for the potential effects of time on depression symptoms.

INTERVENTIONS:
Behavioral: Building Emotion Awareness and Mental Health (BEAM) — The BEAM Program is based on best-practices in telehealth and science-based program design principles aimed at promoting maternal mental health and supportive parenting. The BEAM Program mobile application is designed and managed by Tactica Interactive and hosted on the University of Manitoba secure servers. The weekly group telehealth sessions will be led by clinical coaches (a mental health professional or trainee) and will use the secure videoconferencing platform Zoom (Healthcare license). Parent coaches will be mothers who have recently participated in another research group-based mental health intervention. Parent coaches will engage with participants on the community peer support forum and attend weekly telehealth sessions. The therapeutic aims of the BEAM program are to improve anxiety and depression symptoms and parenting skills using content that draws from the Unified Protocol, and emphasizes self-compassion, effective communication practices, and social support networks.
  Arms: The BEAM program group

SUMMARY:
During the COVID-19 pandemic, the prevalence of maternal depression and anxiety has increased and research suggests that the cognitive development of children born during the pandemic has been impacted. There are significant concerns that a cohort of children may be at-risk for mental illness and impaired self-regulation due to elevated exposure to perinatal maternal mental illness. Intervention is crucial as the intergenerational effects of maternal mental illness are most pronounced when mental health concerns persist. There is currently an urgent need for accessible eHealth interventions for mothers of young children as the pandemic has contributed to an increased prevalence of mental health concerns and to additional barriers to services. The Building Emotion Awareness and Mental Health (BEAM) app-based program was developed to help address maternal mental health concerns and parenting stress. A two-arm randomized controlled trial (RCT) with repeated measures will be used to evaluate the efficacy of the BEAM intervention compared to treatment as usual (TAU) among a sample of 140 mothers who self-report moderate-to-severe symptoms of depression and/or anxiety and have a child 18 to 36 months-old.

DETAILED DESCRIPTION:
Maternal mental health symptoms in the first few years following childbirth are common and can have contributed to adverse consequences for both mother and baby. Two of the most common perinatal mental health concerns are depression and anxiety. The COVID-19 pandemic has introduced heightened stressors for families, including physical isolation from support and social networks, additional childcare responsibilities, and economic uncertainty. Unsurprisingly, the pandemic has also led to an increased prevalence of maternal depression and anxiety in Canada and around the world. These mental health problems are associated with increased health problems and low quality of life for mothers. The COVID-19 pandemic has also posed additional challenges to families and mothers with young children are experiencing heightened parenting stress, increasing their support needs. For mothers with depression, these additional parenting stressors can worsen the symptoms and severity their depression. Furthermore, emerging research suggests that the COVID-19 pandemic has had detrimental effects on early child cognitive development.

According to the developmental origins of health and disease, exposure to maternal depression in the first 5 years of life is linked to children's mental illness, cognitive impairments, and developmental delays. Intervening early is important to help prevent negative long-term consequences for mothers and their children. Without treatment, maternal depressive symptoms tend to remain consistent throughout the preschool years and the adverse consequences of maternal mental health concerns are most pronounced when depression persists. Although there are evidence-based treatments to address maternal mental illness, accessing care can be challenging due to the exceedingly high barriers to service due to COVID-19, such as lack of childcare and time.

Web-based resources have been identified as a preference for mental health support by mothers with mental health problems during the perinatal period. Furthermore, mothers have expressed appreciation for peer support during the perinatal period as social support is often highly relied upon in the postnatal period to care for their infants and themselves. Support from other mothers, specifically, has been found to be helpful in recovering from postpartum depression and individuals report higher satisfaction in treatments of postpartum depression that include a peer support component.

E-health interventions, designed to target both maternal mental illness and parenting abilities, and that prioritize social support, may be a promising avenue to address the intergenerational impact of perinatal mental health problems. The Building Emotion Awareness and Mental Health (BEAM) program is an app-based and online group therapy program that was developed to respond to the high needs of mothers managing depression, anxiety, and parenting stress.

There are 3 objectives for this study:

Evaluate the efficacy of the BEAM app-based program for improving depression compared to a treatment as usual (TAU) control group.

Examine the benefits of BEAM for family relationships, anxiety, parenting stress and behaviours, and child functioning.

Examine exploratory outcomes of parent-child relationship quality, maternal sensitivity, and child emotional reactivity.

ELIGIBILITY:
Inclusion Criteria:

* A mother with a child aged 18-36 months old
* Moderate-to-severe symptoms of depression and/or anxiety (i.e., a score at or above 10 on the Patient Health Questionnaire and/or the General Anxiety Disorder scale
* Comfortable understanding, speaking, and reading English
* Live in Manitoba or Alberta, Canada
* Be available to attend weekly telehealth sessions
* Consent to wearing a Fitbit
* Complete baseline screener and questionnaire and be willing to meet the research team through Zoom (either during assessment or technology check in session).

Exclusion Criteria

* Child is outside of the 18-36 month age range
* Does not meet criteria for moderate-to-severe depression and/or anxiety
* Lives outside of Manitoba or Alberta
* A reported history of attempted suicide in the past year or self-harm in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — "People who identify as mothers"
Enrollment: 140 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change in depression symptoms | The PHQ-9 will be assessed during eligibility screening, pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Symptoms of depression will be assessed using the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a self-administered questionnaire with possible scores ranging from 0 to 27, where higher scores are indicative of more severe symptoms. A cut-off score of ≥ 10 will be used to identify participants who present with clinically concerning symptoms of depression.

SECONDARY OUTCOMES:
Change in parental assistance with child emotion regulation | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Parental assistance with child emotion regulation will be measured using the Parental Assistance with Child Emotion Regulation scale (PACER). The PACER is a parent-report measure of how parents assist children with regulation of emotion using specific strategies. Scores range from 50-350, where higher scores indicate higher engagement in behaviours that support child emotion regulation.
Change in partner social support | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Partner social support will be measured using the Social Support Effectiveness Questionnaire (SSE). The SSE is a self-report measure of partner social support effectiveness .Total scores can range from 0 to 80, with higher scores indicating more effective support.
Change in romantic relationship satisfaction | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Romantic relationship satisfaction will be measured using the 4-item Couple Satisfaction Index (CSI-4). The CSI is a self-report measure of the individual's global evaluations of their romantic relationship. Scores range from 0 to 21, with higher scores reflecting higher levels of satisfaction.
Change in parenting stress | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Parenting stress will be measured using the Parenting Stress Index (PSI), a self-report measure of parenting stress and interactional style across 3 subscales (parent distress, parent-child dysfunction, difficult child) which combine to form a Total Stress scale. Raw scores range from 36 to 180, with higher scores indicating higher levels of parent stress.
Change in parenting discipline practices | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Parenting behaviour and dysfunctional discipline will be measured using the Parenting Scale (PS), a self-rating scale to measure discipline practices in parents of young children. Scores range from 30-210, with higher scores indicating more ineffective parenting discipline practices.
Change in parenting behaviours | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Parenting behaviours will be measured using the Parenting Young Children (PARYC) measure, a self-report of parenting strategies/behaviours relevant for caregivers of young children. Scores range from 21-105, with higher scores indicating more proactive parenting behaviours.
Change in anxiety symptoms | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Maternal anxiety will be measured using the Generalized Anxiety Disorder 7-Item (GAD-7) Scale, a self-rating scale to measure anxiety. Scores range from 0-21, with higher scores indicating higher levels of anxiety.
Change in anger | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Anger will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.1-Anger 5a, a self-report measure to assess the severity and frequency of an individual's anger. Scores range from 5-25, where higher scores indicate more anger.
Change in self-compassion | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Self-compassion will be measured using the Self-Compassion Scale Short-Form (SCS-SF), a self-report measure of self-compassion. Scores range from 12-60, with higher scores indicating higher levels of self-compassion.
Change in sleep problems | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Sleep disturbance will be measured using the PROMIS Sleep Disturbance Scale, a self-report of perceptions of sleep quality, depth, and restoration with the past seven days. Scores range from 8-40, with higher scores indicating greater severity of sleep disturbance.
Change in suicidal ideation severity | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Suicidal ideation severity will be measured using the Depression Symptom Index Suicidality Subscale (DSI-SS), a self-report measure of suicidal ideation. Scores range from 0 to 12, where higher scores indicate higher suicidal ideation.
Change in self-esteem | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Self-esteem will be measured using the Single Item Self-Esteem Scale (SISE), a one-item self-report measure of global self-esteem. Scores range from 1 to 7, where higher scores indicate higher self-esteem.
Change in alcohol use | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Alcohol use will be measured using the Alcohol Use Disorder Identification Test (AUDIT), a self-report measure of alcohol consumption, drinking behaviors, and alcohol-related problems. Scores range from 0 to 40, where higher scores indicate more hazardous alcohol use.
Change in cannabis use | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Cannabis use will be measured using the Cannabis Use Disorder Identification Test - Revised (CUDIT-R), a self-report of cannabis misuse. Scores range from 0 to 32, where higher scores indicate more hazardous cannabis use and scores of 12 or more indicating a possible Cannabis Use Disorder.
Change in child emotional and behavioural problems | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Child emotional and behavioural problems will be measured using the Preschool Pediatric Symptom Checklist (PPSC), a parent report measure of early emotional and behavioural problems in infants and pre-schoolers. Scores range from 0 to 34, where higher scores indicate higher incidence of emotional and behavioural problems
Change in child temperament | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Child temperament will be measured using a subset of questions from the Early Child Behavior Questionnaire (ECBQ), a parent report measure of temperament in children aged 1 to 3. Scores range from 1 to 7, where higher scores indicate higher levels of the temperamental trait.

OTHER OUTCOMES:
Change in parent-child relationship quality | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Parent-child relationship quality will be assessed by coding online video observation
Change in sensitive parenting | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Sensitive parenting will be assessed by coding online video observation
Change in child emotional reactivity | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Child emotional reactivity will be assessed by coding online video observation
Change in heart rate | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Heart rate will be assessed using Fitbit devices
Change in sleep duration | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Sleep duration will be assessed using Fitbit devices
Change in sleep quality | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Sleep quality will be assessed using Fitbit devices
Change in physical activity | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Physical activity will be assessed via step count using Fitbit devices
Feasibility of the BEAM program | To be assessed pre-intervention (T1), immediately after the intervention (T2), and at 6-month follow-up (T3)
  Feasibility of the BEAM program will be assessed using the mHelath App Usability Questionnaire (MAUQ), a self-report measure with three subscales that rate, on a 7-point Likert scale, ease of use (scores range from 5-35), interface and satisfaction (scores range from 7-49), and usefulness (scores range from 6-42), where high scores indicate better useability."

CONTACTS AND LOCATIONS:
Overall Officials: Leslie E Roos, PhD, Principal Investigator — University of Manitoba; Lianne Tomfohr-Madsen, PhD, Principal Investigator — University of Calgary
Locations (1):
- The University of Manitoba - Department of Psychology, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data (e.g. standardized questionnaire responses, aggregated program use data, sociodemographics linked to an identifier number) may be made available on public data platforms such as open science framework or a requirement by a granting agency or journal.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Xie EB, Simpson KM, Reynolds KA, Giuliano RJ, Protudjer JLP, Soderstrom M, Sauer-Zavala S, Giesbrecht GF, Lebel C, Mackinnon AL, Rioux C, Penner-Goeke L, Freeman M, Salisbury MR, Tomfohr-Madsen L, Roos LE. Building Emotional Awareness and Mental Health (BEAM): study protocol for a phase III randomized controlled trial of the BEAM app-based program for mothers of children 18-36 months. Trials. 2022 Sep 5;23(1):741. doi: 10.1186/s13063-022-06512-5. PMID 36064436